CLINICAL TRIAL: NCT03453567
Title: Evaluation of Effectiveness and Safety of Aortic Valve Replacement in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of Aortic Valve Replacement in Routine Clinical Practice
Acronym: IRIS AVR
Status: Active, not recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2018-04
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis
Keywords: TAVR; SAVR; TAVI; Conventional AVR; Sutureless AVR
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TAVR: Transcatheter Aortic Valve Replacement
  Interventions: Procedure: Valve Replacement
- Sutureless AVR: Sutureless Aortic Valve Replacement
  Interventions: Procedure: Valve Replacement
- Conventional AVR: Conventional Aortic Valve Replacement
  Interventions: Procedure: Valve Replacement

INTERVENTIONS:
Procedure: Valve Replacement — Aortic valve replacement

SUMMARY:
This study evaluated effectiveness and safety of aortic valve replacement in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Patient with aortic valve replacement

Exclusion Criteria:

* Combined with mitral stenosis requiring surgery or aorta stenosis
* Acute bacterial endocarditis within 1 month of valve replacement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve replacement
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 1 year

SECONDARY OUTCOMES:
Cardiovascular mortality | 5 years
  A. Death due to proximate cardiac cause B. Death caused by noncoronary vascular condition C. All procedure-related/surgery-related death D. All valve-related death E. Sudden or unwitnessed death F. Death of unknown cause
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Myocardial infarction | 5 years
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
All stroke and transient ischemic attack | 5 years
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Bleeding | 5 years
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Access site complication | 5 years
  Operation site complication Vascular access site and access-related complication
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Acute kidney injury | 5 years
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Permanent pacemaker insertion | 5 years
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
TAVR-related complication | 5 years
  A. Conversion to open surgery B. Coronary obstruction C. Mitral valve apparatus damage or dysfunction D. Cardiac tamponade E. Endocarditis F. Valve thrombosis G. Valve malpositioning H. TAV-in-TAV deployment
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Prosthetic valve dysfunction | 5 years
  A. Prosthetic aortic valve stenosis B. Prosthesis-patient mismatch C. Prosthetic aortic valve regurgitation
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Composite event | 5 years
  A. Device success B. Early safety (30 days)
  * Death, stroke, life-threatening bleeding, acute kidney injury, coronary stenosis requiring intervention, significant vascular complication, valve dysfunction requiring intervention C. Clinical efficacy (30 days)
  * Death, stroke, deteriorating heart failure or valve function requiring hospitalization, NYHA III or IV dyspnea, valve dysfunction
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
Structural valve deterioration | 5 years
  Either Discharge or 30-day, at the earliest time point
  1-,6-, and 12-months, and 3-,5-years
NYHA class | 30 days and 1 year
  New York Heart Association (NYHA) Functional Classification
The change of valve area | 30 days and 1 year
  Aortic valve area measured by echocardiography (mm2)
New onset atrial fibrillation | 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Jung Choo, MD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Sejong Hospital, Bucheon-si
  - Asan Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided